CLINICAL TRIAL: NCT06836037
Title: A Single and Multiple Dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics of MK-6024 in Healthy Chinese Participants
Brief Title: A Clinical Study of Efinopegdutide (MK-6024) in Healthy Chinese Volunteers (MK-6024-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6024-011; MK-6024-011 (Other: MSD); 2020-005136-30 (Registry Identifier: EU CT)
Record Dates: First submitted 2025-02-18; First posted 2025-02-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Efinopegdutide Low Dose (Experimental): Participants receive low dose efinopegdutide at a single dose on day 1
  Interventions: Drug: Efinopegdutide
- Efinopegdutide Medium dose (Experimental): Participants receive medium dose efinopegdutide at a single dose on day 1
  Interventions: Drug: Efinopegdutide
- Efinopegdutide High Dose (Experimental): Participants receive high dose efinopegdutide at a single dose on day 1
  Interventions: Drug: Efinopegdutide
- Efinopegdutide Multiple Dose (Experimental): Participants receive multiple doses of efinopegdutide over 78 days
  Interventions: Drug: Efinopegdutide
- Placebo (Placebo Comparator): Participants receive placebo to match efinopegdutide dose and regimen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efinopegdutide — Subcutaneous injection
  Other Names: MK-6024; HM12525A; JNJ-64565111,
  Arms: Efinopegdutide High Dose; Efinopegdutide Low Dose; Efinopegdutide Medium dose; Efinopegdutide Multiple Dose
Drug: Placebo — placebo matching efinopegdutide
  Arms: Placebo

SUMMARY:
The goal of this study is to learn about the safety and whether people tolerate a study medicine called efinopegdutide. The study will also measure what happens to efinopegdutide in a healthy person's body over time.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥25 and ≤35 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Had major surgery, donated or lost approximately 400 mL blood within 4 weeks prior to entering the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 112 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 78 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Maximum Plasma Concentration (Cmax) of Efinopegdutide- single dose | At designated time points up to 35 days
  Blood samples will be collected to determine the Cmax of efinopegdutide when administered as a single dose
Time to Maximum Plasma Concentration (Tmax) of Efinopegdutide- single dose | At designated time points up to 35 days
  Blood samples will be collected to determine the Tmax of efinopegdutide when administered as a single dose
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Efinopegdutide- single dose | At designated timepoints up to 35 days
  Blood samples will be collected to determine the AUC0-last of efinopegdutide when administered as a single dose
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) of Efinopegdutide- single dose | At designated timepoints up to 35 days
  Blood samples will be collected to determine the AUC0-inf of efinopegdutide when administered as a single dose
Terminal half life (t1/2) of Efinopegdutide- single dose | At designated timepoints up to 35 days
  Blood samples will be collected to determine the t1/2 of efinopegdutide when administered as a single dose
Apparent Clearance (CL) of Efinopegdutide- single dose | At designated timepoints up to 35 days
  Blood samples will be collected to determine the CL of efinopegdutide when administered as a single dose
Volume of Distribution (Vz) of Efinopegdutide- single dose | At designated timepoints up to 35 days
  Blood samples will be collected to determine the Vz of efinopegdutide when administered as a single dose
Maximum Plasma Concentration (Cmax) of Efinopegdutide- multiple dose | At designated time points up to 112 days
  Blood samples will be collected to determine the Cmax of efinopegdutide when multiple doses are administered
Minimum Plasma Concentration (Cmin) of Efinopegdutide- multiple dose | At designated time points up to 112 days
  Blood samples will be collected to determine the Cmin of efinopegdutide when multiple doses are administered
Time to Maximum Plasma Concentration (Tmax) of Efinopegdutide- multiple dose | At designated time points up to 112 days
  Blood samples will be collected to determine the Tmax of efinopegdutide when multiple doses are administered
Terminal half life (t1/2) of Efinopegdutide- multiple dose | At designated timepoints up to 112 days
  Blood samples will be collected to determine the t1/2 of efinopegdutide when multiple doses are administered
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Efinopegdutide-multiple dose | At designated timepoints up to 112 days
  Blood samples will be collected to determine the AUC0-last of efinopegdutide when multiple doses are administered
Apparent Clearance (CL) of Efinopegdutide- multiple dose | At designated timepoints up to 112 days
  Blood samples will be collected to determine the CL of efinopegdutide when multiple doses are administered
Volume of Distribution at Steady State (Vss) of Efinopegdutide- multiple dose | At designated timepoints up to 112 days
  Blood samples will be collected to determine the Vss of efinopegdutide when multiple doses are administered
Area Under the Concentration-Time Curve to the end of the dosing period (AUC 0-tau)of Efinopegdutide- multiple dose | At designated timepoints up to 78 days
  Blood samples will be collected to determine the AUC0 to tau of efinopegdutide when multiple doses are administered

SECONDARY OUTCOMES:
Change from Baseline in Weight | Baseline and day 112
  Change from baseline in weight will be computed for participants who received multiple doses of efinopegdutide
Change from Baseline in HDL Cholesterol | Baseline and day 112
  Change from baseline in HDL cholesterol will be computed for participants who received multiple doses of efinopegdutide
Change from Baseline in LDL Cholesterol | Baseline and day 112
  Change from baseline in LDL cholesterol will be computed for participants who received multiple doses of efinopegdutide
Change from Baseline in Total Cholesterol | Baseline and day 112
  Change from baseline in total cholesterol will be computed for participants who received multiple doses of efinopegdutide
Change from Baseline in Triglycerides | Baseline and day 112
  Change from baseline in triglycerides will be computed for participants who received multiple doses of efinopegdutide
Number of participants with anti drug antibodies (ADA) to efinopegdutide | At designated timepoints up to 112 days
  Blood samples will be collected to determine the number of participants with ADA to efinopegdutide

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Zhongshan Hospital,Fudan University-Dep. of Clinical Pharmacology (Site 0001), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com